CLINICAL TRIAL: NCT03403088
Title: Non-carious Cervical Lesions: Clinical Comparison of Different Strategies to Treat Dentin Hypersensitivity
Brief Title: Non-carious Cervical Lesions and Treatments
Acronym: NCCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Camila Tirapelli, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04969312.6.0000.5419
Record Dates: First submitted 2018-01-02; First posted 2018-01-18 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Tooth Sensitivity
Keywords: Non-carious cervical lesions; dentin hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Low-Level Light Therapy; Resin Cements

STUDY DESIGN:
Intervention Model Description: 60 participants with NCCLs and positive for DH are enrolled in the study to receive randomly the followed treatments: LA= 780 nm and 70mW GaAlAs Laser/ 4 sessions; LAP= placebo laser/ four sessions; CP= ClinproTM XT Varnish/ in-office single session; RX= adhesive RelyXTM Arc/ in-office single session; DE= stannous fluoride dentifrice/30-days-home-use; DE-P= placebo dentifrice/30-days-home-use
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group LA (Experimental): INTERVENTION: to apply Laser (780 nm and 70mW) at the cementum-enamel junction fat the teeth affected by sensitivity
  Interventions: Device: Experimental: • Group LA
- Group LA-P (Placebo Comparator): INTERVENTION: to apply Laser (780 nm and 70mW) at the cementum-enamel junction at the teeth affected by sensitivity with the laser device having no effective laser emission, only guided by light
  Interventions: Device: Placebo Comparator: • Group LA-P
- Group DE (Experimental): INTERVENTION: to brush teeth with a blinded dentifrice with 0,45% of stannous fluoride and a soft-bristled manual toothbrush (Johnson & Johnson®).
  Interventions: Other: Experimental: • Group DE
- Group DE-P (Placebo Comparator): INTERVENTION: to brush teeth with a blinded dentifrice with 1500 ppm of available fluoride and a soft-bristled manual toothbrush (Johnson & Johnson®).
  Interventions: Other: Placebo Comparator: • Group DE-P
- Group RGI (Experimental): INTERVENTION: to apply a thin layer of resin based glass-ionomer product on the cervical surface of the affected teeth affected by sensitivity following the manufacturer instructions.
  Interventions: Other: Experimental: • Group RGI
- Group RX (Experimental): INTERVENTION: to apply Adper Single Bond Plus Adhesive in accordance with the manufacturer instructions, at the teeth affected by sensitivity
  Interventions: Other: Experimental: Group RX

INTERVENTIONS:
Device: Experimental: • Group LA — to apply Laser (780 nm and 70mW) at the cementum-enamel junction fat the teeth affected by sensitivity
  Other Names: low laser therapy
  Arms: Group LA
Device: Placebo Comparator: • Group LA-P — to apply Laser (780 nm and 70mW) at the cementum-enamel junction at the teeth affected by sensitivity with the laser device having no effective laser emission, only guided by light
  Other Names: low laser therapy
  Arms: Group LA-P
Other: Experimental: • Group DE — to brush teeth with a blinded dentifrice with 0,45% of stannous fluoride and a soft-bristled manual toothbrush (Johnson & Johnson®).
  Other Names: desensitizing dentifrice
  Arms: Group DE
Other: Placebo Comparator: • Group DE-P — to brush teeth with a blinded dentifrice with 1500 ppm of available fluoride and a soft-bristled manual toothbrush (Johnson & Johnson®).
  Other Names: placebo desensitizing dentifrice
  Arms: Group DE-P
Other: Experimental: • Group RGI — to apply a thin layer of resin based glass-ionomer product on the cervical surface of the affected teeth affected by sensitivity following the manufacturer instructions.
  Other Names: resin glass ionomer restorarion
  Arms: Group RGI
Other: Experimental: Group RX — to apply Adper Single Bond Plus Adhesive in accordance with the manufacturer instructions, at the teeth affected by sensitivity product for 20 seconds.
  Other Names: selant with resin cement
  Arms: Group RX

SUMMARY:
This study will compare clinically the efficacy, time to action and duration of different treatments for patients with non-carious cervical lesions (NCCLs) that caused dentin hypersensitivity (DH).

DETAILED DESCRIPTION:
This study will compare clinically the efficacy, time to action and duration of different treatments for patients with non-carious cervical lesions (NCCLs) that caused dentin hypersensitivity (DH). Casuistic and methods: 60 participants with NCCLs and positive for DH will be enrolled in the study to receive randomly the followed treatments: LA= 780 nm and 70mW GaAlAs Laser/ 4 sessions; LAP= placebo laser/ four sessions; RGI= ClinproTM XT Varnish/ in-office single session; RX= adhesive RelyXTM Arc/ in-office single session; DE= stannous fluoride dentifrice/30-days-home-use; DE-P= placebo dentifrice/30-days-home-use. Pain from DH is measured with visual analogue scale (VAS), pre-treatment and in accordance with each treatment, immediately after the end of the treatment (S1); one and two weeks (1S and 2S) and one and two months (1M and 2M) after the end of the treatments. Strategies of treatments are compared each other in each period of evaluation and along time with pre-treatments values of pain, using Kruskall-Wallis and Friedman Test (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

- (a) male or female between 18 to 60 years old; (b) good general (no diseases that could interfere in the results) and oral health (no alterations in hard or soft tissues); (c) a minimum of 24 permanent teeth; (d) presence of non-carious cervical lesion; and (e) compliment of cervical dentin hypersensitivity

Exclusion Criteria:

-(a) chronic analgesic or anti-inflammatory therapy; (b) orthodontic treatment or dental prosthesis; (c) desensitization therapy in the preceding 3 months; (d) alimentary disorder or acid diet; and (e) pregnant or lactating women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
pain from dentin hypersensitivity (DH) | pre-treatment
  Examiner assess dentin hypersensitivity (DH) using VAS (visual analogue scale). The selected tooth was thermic stimulated by a cold air (approximately 10°C) from a triple syringe placed 3mm from the buccal surface in the cervical area, perpendicular to the tooth long axis at full blast during 3 seconds. In addition, the selected tooth received a mechanical stimulus by a dental probe n° 05 over the cervical area. Thereby, volunteers were instructed to record the sensitivity perception by placing a mark on the scale from 0 (no pain) to 10 (intolerable pain) while sensitivity test was occurred
pain from dentin hypersensitivity (DH) | immediately after the end of the treatment (S1);
  Examiner assess dentin hypersensitivity (DH) using VAS (visual analogue scale). The selected tooth was thermic stimulated by a cold air (approximately 10°C) from a triple syringe placed 3mm from the buccal surface in the cervical area, perpendicular to the tooth long axis at full blast during 3 seconds. In addition, the selected tooth received a mechanical stimulus by a dental probe n° 05 over the cervical area. Thereby, volunteers were instructed to record the sensitivity perception by placing a mark on the scale from 0 (no pain) to 10 (intolerable pain) while sensitivity test was occurred
pain from dentin hypersensitivity (DH) | one weeks (1S) after the end of the treatments
  Examiner assess dentin hypersensitivity (DH) using VAS (visual analogue scale). The selected tooth was thermic stimulated by a cold air (approximately 10°C) from a triple syringe placed 3mm from the buccal surface in the cervical area, perpendicular to the tooth long axis at full blast during 3 seconds. In addition, the selected tooth received a mechanical stimulus by a dental probe n° 05 over the cervical area. Thereby, volunteers were instructed to record the sensitivity perception by placing a mark on the scale from 0 (no pain) to 10 (intolerable pain) while sensitivity test was occurred
pain from dentin hypersensitivity (DH) | two weeks (2S) after the end of the treatments
  Examiner assess dentin hypersensitivity (DH) using VAS (visual analogue scale). The selected tooth was thermic stimulated by a cold air (approximately 10°C) from a triple syringe placed 3mm from the buccal surface in the cervical area, perpendicular to the tooth long axis at full blast during 3 seconds. In addition, the selected tooth received a mechanical stimulus by a dental probe n° 05 over the cervical area. Thereby, volunteers were instructed to record the sensitivity perception by placing a mark on the scale from 0 (no pain) to 10 (intolerable pain) while sensitivity test was occurred
pain from dentin hypersensitivity (DH) | One month (1M) after the end of the treatments
  Examiner assess dentin hypersensitivity (DH) using VAS (visual analogue scale). The selected tooth was thermic stimulated by a cold air (approximately 10°C) from a triple syringe placed 3mm from the buccal surface in the cervical area, perpendicular to the tooth long axis at full blast during 3 seconds. In addition, the selected tooth received a mechanical stimulus by a dental probe n° 05 over the cervical area. Thereby, volunteers were instructed to record the sensitivity perception by placing a mark on the scale from 0 (no pain) to 10 (intolerable pain) while sensitivity test was occurred
pain from dentin hypersensitivity (DH) | Two months (2M) after the end of the treatments
  Examiner assess dentin hypersensitivity (DH) using VAS (visual analogue scale). The selected tooth was thermic stimulated by a cold air (approximately 10°C) from a triple syringe placed 3mm from the buccal surface in the cervical area, perpendicular to the tooth long axis at full blast during 3 seconds. In addition, the selected tooth received a mechanical stimulus by a dental probe n° 05 over the cervical area. Thereby, volunteers were instructed to record the sensitivity perception by placing a mark on the scale from 0 (no pain) to 10 (intolerable pain) while sensitivity test was occurred

CONTACTS AND LOCATIONS:
Overall Officials: Takami Hirono Hotta, PhD, Study Director — USP
Locations (1):
- University of Sao Paulo -Ribeirao Preto Campus, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) available to other researchers will be not available for other researchers